CLINICAL TRIAL: NCT07301281
Title: Cluster Randomized Controlled Trial of the "Mittin" Intervention in Addis Ababa, Ethiopia
Brief Title: Trial of the "Mittin" Intervention to Improve Contraceptive Side Effect Counseling and Follow-up in Ethiopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: St. Paul's Hospital Millennium Medical College, Ethiopia (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 24-43085; INV-044992 (Other Grant/Funding Number: Gates Foundation)
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Contraception; Side Effects

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Arm will be masked to the principal investigators until analysis of the primary outcomes at 4 months; prior to this data will be in aggregate form and will not reveal intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care arm (No Intervention): Health centers randomized to the standard of care arm will continue offering standard of care contraceptive counseling as per Ethiopian Ministry of Health guidelines. After completion of the c-RCT, the control arm health centers will receive Mittin materials for use on-site (counseling tools, waiting room posters, and educational handouts).
- Mittin Intervention arm (Experimental): Health centers randomized to receive the Mittin intervention will receive staff training and materials (counseling tools, waiting room posters, and educational handouts) necessary to offer Mittin's side effects counseling and support model in their facilities. Women enrolled in the study in intervention health centers will receive proactive follow-up calls from call center agents to offer support after initiating a new contraceptive method. The call center will also be available on-demand to any person who desires support related to contraceptive options or side effects.
  Interventions: Behavioral: Mittin

INTERVENTIONS:
Behavioral: Mittin — Mittin intervention consists of the following components:
  1. Educational posters and handouts to raise awareness of the right to contraceptive choice and to switch methods if side effects become intolerable
  2. Decision support tools for providers to aid women in weighing the risks and benefits of potential side effects during in-person counseling
  3. On-demand and proactive virtual side effects counseling and referrals via a call center.
  Arms: Mittin Intervention arm

SUMMARY:
The goal of this clinical trial is to learn if the "Mittin" intervention can improve women's ability to manage their fertility in line with their preferences among women aged 15-49 using hormonal contraceptives or intrauterine devices and attending public health centers in Addis Ababa, Ethiopia. The main question it aims to answer is: Does the Mittin intervention increase preference-aligned fertility management, contraceptive method satisfaction, and preferred contraceptive method use among participants compared to standard care?

Researchers will compare women's outcomes in health centers providing the Mittin intervention to women's outcomes in health centers that offer standard care to see if Mittin improves women's ability to act in line with their contraceptive preferences.

Participants will

* Receive either standard contraception services (control arm) or enhanced services (intervention arm)
* Participate in a survey at the beginning of the study
* Participate in surveys 4 and 8 months later

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Started or continued using hormonal contraceptive method or copper IUD on day of recruitment
* Ages 15-49 years
* Willing to provide phone number and receive follow-up phone call

Exclusion Criteria:

* Not planning to live in Addis Ababa for the next eight months
* Can not verbally communicate
* Not willing to provide consent for the study

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2715 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Preference-Aligned Fertility Management (PFM) Index | Measured at 4 and 8 months
  The PFM Index measures whether use or non-use of contraception aligns with one's preferences. It is a binary measure where 0=no alignment, and 1=alignment.

SECONDARY OUTCOMES:
Agency in Contraceptive Decisions Scale | Measured at 4 and 8 months
  This 15-item scale includes individual items scored on a scale 0-3. The composite score is an average of scores on all items. 3=highest agency.
Method satisfaction | Measured at 4- and 8-months
  1-item measure where 1=very dissatisfied and 5=very satisfied
Preferred Method Use | Measured at 4 and 8 months
  Single item assesses whether there is a contraceptive method that a person would like to use but is not currently using (Yes/No/Uncertain)

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Holt, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- St. Paul's Hospital Millennium Medical College, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
No later than six months after publication of the initial findings of the study, we will make individual participant data that underlie the results available in a public repository after deidentification.
Time Frame: Within 6 months of publication of findings, with no end date
Access Criteria: Anyone will be able to access publicly available deidentified data once it is uploaded to a repository.